CLINICAL TRIAL: NCT05769985
Title: Study on the Interaction Between Psychological States and Caregiver's Responses on Pain in Patients Suffering From Chronic Pain
Brief Title: Interaction Between Psychological States and Caregiver's Responses on Pain in Patients Suffering From Chronic Pain
Acronym: CARE-ME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 03C213
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Caregiver's responses and patient satisfaction — Interaction between caregivers' responses and patient satisfaction about those responses

SUMMARY:
Chronic pain is a major cause of disability, and given its negative impact on the functional, psychological, and social well-being of sufferers, it is crucial to identify the biopsychosocial factors that influence it. While biological and psychological factors have been extensively studied, the role of the patient's relational context has not been thoroughly investigated to date. The presence of pain affects both directly and indirectly the patient's family and social context, which could significantly influence the perception of pain itself. In particular, partners of chronic pain patients may experience high levels of stress, anxiety, and worry, and this may have an impact on couple satisfaction and the type of partner's responses with respect to the patient's pain manifestations. It is conceivable that the type of interaction between patient and partner is influenced by the intersection of the ways in which the patient expresses pain, such as by manifesting catastrophic experiences, with the type of responses provided by the partner, such as of criticism, distraction, or support. It can be hypothesized that both the partner's actual responses to the patient's manifestations of pain and the patient's satisfaction with these responses are important. This study therefore aims to understand the relationships between these factors. Specifically, it will assess whether attributions and catastrophizing behaviors of the patient influence pain intensity and interference over time through mediation by the responses given by the partner. It will also be assessed whether this mediation is moderated by the patient's satisfaction with the partner's responses.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of condition associated with chronic pain
* Presence of a caregiver associated by kinship and living together for at least six months
* Having given written consent at the time of treatment received at one of the OUs involved in the project to the possibility of being contacted to participate in research for scientific purposes.

Exclusion Criteria:

* Patients diagnosed with psychosis, dementia, or psychiatric comorbidities
* Patients who, at the time of recruitment, will be hospitalized or who will be undergoing inpatient rehabilitation treatment or who will have a scheduled surgery to be performed during the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 7 days
  Pain intensity as measured by a 0-10 Numeric Rating Scale
Pain interference | 7 days
  Pain interference as measured by a 0-10 Numeric Rating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Auxologico Mosè Bianchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be uploaded to an online repository